CLINICAL TRIAL: NCT07102524
Title: A Phase 1/2 Open-Label Intrathecal Administration of TSHA-105 to Determine the Safety and Efficacy in 2 Subjects With SLC13A5 Citrate Transporter Disorder Caused by a Mutation in the SLC13A5 Gene
Brief Title: Intrathecal Gene Therapy For SLC13A5 Citrate Transporter Disorder
Acronym: SLC13A5
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TESS Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLC13A5 Gene Therapy; AAV9/SLC13A5 (Other: TSHA-105)
Record Dates: First submitted 2025-07-21; First posted 2025-08-03 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: SLC13A5 Citrate Transporter Disorder
Keywords: SLC13A5; AAV9; Epileptic Encephalopathy; SLC13A5 Deficiency; SLC13A5 Citrate Transporter Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TSHA-105 treament (Experimental): TSHA-105 Treatment
  Interventions: Drug: TSHA-105

INTERVENTIONS:
Drug: TSHA-105 — AAV9/SLC13A5

SUMMARY:
Phase 1/2, open-label study to assess the efficacy and safety of a single lumbar intrathecal administration of TSHA-105 in individuals with SLC13A5 Citrate Transporter Disorder

DETAILED DESCRIPTION:
TSHA-105 is an AAV9-based gene therapy vector that expresses the fully functional form of SLC13A5 under the control of a synthetic promoter. TSHA-105 will be delivered intrathecally and is designed to achieve stable, potentially life-long expression of SLC13A5 protein in non-dividing cells. This clinical study is a pivotal open-label phase 1/2 study designed to assess safety and efficacy of TSHA-105 in individuals with SLC13A5 Citrate Transporter Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and females between the ages of 2 to 9 and 10 to 20 years at the time of screening
* Confirmed diagnosis of SLC13A5 citrate transporter disorder by genomic DNA mutation analysis demonstrating homozygous or compound heterozygous, confirmed pathogenic variants in the SLC13A5 gene
* Clinical features consistent with SLC13A5 citrate transporter disorder
* Written informed consent provided by subject/parent/guardian and willingness to participate and comply with all the study related visits and procedures. Assent provided by children 10 to 17 years old based on their ability to understand the risks and possible benefits, and the activities expected of them.
* Subjects able to reproduce must use a barrier method of contraception for the first 12 months after dosing as well as at least one additional highly effective birth control method if sexually active

Exclusion Criteria:

* Inability to participate in study procedures (as determined by the site investigator)
* Presence of a concomitant medical condition that precludes lumbar puncture (LP) or use of anesthetics
* History of bleeding disorder or any other medical condition or circumstance in which lumbar puncture is contraindicated according to local institutional policy
* Inability to be safely sedated in the opinion of the clinical anesthesiologist
* Active infection, at the time of dosing, based on clinical observations
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer
* Inability of the subject to undergo MRI according to local institutional policy
* Inability of the subject to undergo any other procedure required in this study
* The presence of significant non-SLC13A5 related CNS impairment or behavioral disturbances that would confound the scientific rigor or interpretation of results of the study
* Have received an investigational drug within 30 days prior to screening or plan to receive an investigational drug (other than gene therapy) during the study.
* Enrollment and participation in another interventional clinical trial
* Contraindication to TSHA-105 or any of its ingredients
* Contraindication to any of the immune suppression medications used in this study
* Clinically significant abnormal laboratory values (hemoglobin < 6 or > 20 g/dL; white blood cell > 20,000 per cmm, platelets count < 100,000 per cmm; INR > ULN; GGT, ALT, and AST or total bilirubin > 2x ULN, creatinine ≥ 1.5 mg/dL) prior to gene replacement therapy

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 5 years
  Safety measured by:
  * Incidence of AEs/SAEs considered related to TSHA-105 and grade 3 or higher as per the Common Terminology Criteria for Adverse Events through month 24
  * Clinical Safety Labs (Chemistry, Hematology, Coagulation, Lipids, Cardiac Safety, Urinalysis), Vital Signs, EKGs, Trans-thoracic Echocardiogram

SECONDARY OUTCOMES:
Peabody Developmental Motor Scales, 2nd Edition | 5 Years
  Assesses fine and gross motor skills in children from birth to 5 years.
  Subtests include reflexes, locomotion, object manipulation, grasping, and visual-motor integration.
Mullens Scales of Early Learning | 5 Years
  Evaluates cognitive and motor development in children from birth to 68 months.
  Measures visual reception, fine motor, expressive language, and receptive language.
SLC13A5 Deficiency Movement Assessment Scale | 5 years
  A disease-specific tool developed to evaluate motor function and movement abnormalities in children with SLC13A5 deficiency
Vineland Adaptive Behavior Scale, 3rd Edition | 5 years
  Measures adaptive behaviors including communication, daily living skills, socialization, and motor skills.
PedsQL Family Impact Module | 5 years
  Measures the impact of pediatric chronic health conditions on parents and families.
  Focuses on emotional, social, and cognitive functioning, as well as communication and worry.
PedsQL Epilepsy Module | 5 Years
  A disease-specific quality-of-life tool designed for children with epilepsy.
  Assesses cognitive functioning, worry, impact, and communication.
Seizure Diary | 5 years
  A caregiver-completed log for tracking seizure frequency, duration, type, and possible triggers.
  For evaluating treatment response and seizure patterns.
Physician Clinical Global Impression (CGI) | 5 years
  A clinician-rated scale that evaluates illness severity and improvement over time.
Parent-Assessed Clinical Global Impression (PGI) | 5 years
  A caregiver's subjective assessment of the child's overall functioning and response to treatment
Sleep Disturbance Scale for Children | 5 years
  A parent-reported tool for assessing sleep problems in children aged 6.5-15 years.
  Evaluates disorders like insomnia, sleep-disordered breathing, and excessive somnolence

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Essential documents
Supporting Information: Study Protocol
Time Frame: 5 years